CLINICAL TRIAL: NCT00284934
Title: A Multicenter, National, Open-label, Prospective, Randomized Study to Evaluate Efficacy and Tolerability of Enteric-coated Mycophenolate Sodium 1440 mg/Day With Tacrolimus Reduced Dose Versus Enteric-coated Mycophenolate Sodium 720 mg/Day With Tacrolimus Standard Dose, in Maintenance, Stable, Adult, Kidney Transplant Recipients
Brief Title: Enteric-coated Mycophenolate Sodium (EC-MPS) With Reduced-dose Tacrolimus Versus EC-MPS With Standard-dose Tacrolimus in Stable Kidney Transplant Recipients
Acronym: OLYMPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AFR04
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-03

CONDITIONS: Kidney Diseases
Keywords: Dose optimization; immune suppressive regimen; enteric-coated mycophenolate sodium; EC-MPS; renal transplantation; kidney; transplant; maintenance patients; Renal transplantation in maintenance
MeSH Terms: conditions — Kidney Diseases | interventions — Mycophenolic Acid; Tacrolimus; Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dose EC-MPS (Active Comparator): Patients received 720 mg/day (360 mg twice a day (bid) orally) Enteric-coated mycophenolate sodium (EC-MPS) and tacrolimus dose (twice a day orally) adjusted to maintain the trough blood level (C0) contained between 5.5 and 10 ng/mL. The randomization was stratified on 1 factor: treatment with or without steroids. Prednisone (or oral equivalent) was administrated to patients as before entering the study and as per center's standard practice, but at a dose of at least 5 mg/day.
  Interventions: Drug: Enteric-coated mycophenolate sodium (EC-MPS); Drug: Tacrolimus; Drug: Corticosteroids
- High EC-MPS (Experimental): Patients received 1440 mg/day (720 mg twice a day (bid) orally) Enteric-coated mycophenolate sodium (EC-MPS) and tacrolimus dose (twice a day orally) tapered to reach a trough blood level target contained between 2 and 4.5 ng/mL within 15 days after randomization at the most. The randomization was stratified on 1 factor: treatment with or without steroids. Prednisone (or oral equivalent) was administrated to patients as before entering the study and as per center's standard practice, but at a dose of at least 5 mg/day.
  Interventions: Drug: Enteric-coated mycophenolate sodium (EC-MPS); Drug: Tacrolimus; Drug: Corticosteroids

INTERVENTIONS:
Drug: Enteric-coated mycophenolate sodium (EC-MPS)
  Other Names: Myfortic
Drug: Tacrolimus
  Other Names: Prograf
Drug: Corticosteroids — At a dose of at least 5 mg/day.
  Other Names: Prednisone

SUMMARY:
This study introduces a new optimization immunosuppressive regimen associating tacrolimus at a reduced dose and enteric-coated mycophenolate sodium at an increased dose in order to slow down renal function worsening and to prevent the progression of chronic allograft nephropathy, while maintaining the same efficacy, in maintenance renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary kidney transplant
* Treatment with mycophenolic acid (MMF 1 g/d or EC-MPS 720 mg/d) and tacrolimus (trough concentration [C0] ≥ 5.5 ng/mL)
* Creatinine clearance ≥ 30 mL/min and < 60 mL/min and stable renal function

Exclusion Criteria:

* Multi-organ recipients or previous transplant with any other organ different from kidney
* Biopsy proven acute rejection or treated acute rejection within the last 3 months.
* Prescription of mycophenolate mofetil 1 g/d or mycophenolate sodium 720 mg/d due to adverse event occurrence when higher doses were administered

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Derived] Kamar N, Rostaing L, Cassuto E, Villemain F, Moal MC, Ladriere M, Barrou B, Ducloux D, Chaouche K, Quere S, Di Giambattista F, Be F. A multicenter, randomized trial of increased mycophenolic acid dose using enteric-coated mycophenolate sodium with reduced tacrolimus exposure in maintenance kidney transplant recipients. Clin Nephrol. 2012 Feb;77(2):126-36. doi: 10.5414/CN107227. PMID 22257543

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Dose EC-MPS: Patients received 720 mg/day (360 mg twice a day (bid) orally) Enteric-coated mycophenolate sodium (EC-MPS) and tacrolimus (twice a day orally) dose adjusted to maintain a trough blood level (C0) between 5.5 and 10 ng/mL. The randomization was stratified on 1 factor: treatment with or without steroids. Prednisone (or oral equivalent) was administrated to patients as before entering the study and as per center's standard practice, but at a dose of at least 5 mg/day.
- High EC-MPS: Patients received 1440 mg/day (720 mg twice a day orally) Enteric-coated mycophenolate sodium (EC-MPS) and tacrolimus (twice a day orally) dose tapered to reach a trough blood level target of between 2 and 4.5 ng/mL within 15 days after randomization. The randomization was stratified on 1 factor: treatment with or without steroids. Prednisone (or oral equivalent) was administrated to patients as before entering the study and as per center's standard practice, but at a dose of at least 5 mg/day.
Period: Overall Study
Arm/Group | Standard Dose EC-MPS | High EC-MPS
Started | 48 | 46
Intent-to-treat Population (ITT) | 47 | 45
Completed | 44 | 43
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Other reasons | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose EC-MPS | High EC-MPS | Total
Number analyzed (Participants) | 47 | 45 | 92
Age Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (10.4) | 50.7 (12.2) | 52.7 (11)
Age, Customized [Number; unit: Participants]
  < 45 | 11 | 13 | 24
  45-60 | 18 | 20 | 38
  >= 60 | 18 | 12 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Renal Function Assessed by Change in Estimated Glomerular Filtration Rate(eGFR)
Description: Change in estimated glomerular filtration rate from baseline to Month 6 calculated by using abbreviated Modification of Diet in Renal Disease (MDRD) formula. Modification of Diet in Renal Disease (MDRD) formula is: GFR [mL/min/1.73m^2] = 186.3*(C^-1.154)*(A^-0.203)*G*R where -C is the serum concentration of creatinine [mg/dL], -A is patient age at sample collection date [years], -G=0.742 when gender is female, otherwise G=1, -R=1.21 when race is black, otherwise R=1.
Time Frame: Baseline and Month 6
Population: Intent-to-treat (ITT) population was defined as all patients who were randomized and treated with study medication and had at least one post-treatment efficacy assessment.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Standard Dose EC-MPS | High EC-MPS
Number analyzed (Participants) | 47 | 45
mL/min/1.73m^2
  Baseline (n= 47, 45) | 45.3 (9.5) | 56.4 (11.2)
  Month 6 (n= 45, 43) | 44.7 (11.5) | 49.1 (11.11)
  Change from Baseline - Month 6 (n= 45, 43) | -0.4 (6.9) | 2.4 (6.1)

2. Secondary Outcome: Renal Function at 3 Months Assessed by Change in Estimated Glomerular Filtration Rate (eGFR)
Description: Change in estimated glomerular filtration rate from baseline to Month 3 calculated by using abbreviated MDRD formula. Modification of Diet in Renal Disease (MDRD) formula is: GFR [mL/min/1.73m^2] = 186.3*(C^-1.154)*(A^-0.203)*G*R where -C is the serum concentration of creatinine [mg/dL], -A is patient age at sample collection date [years], -G=0.742 when gender is female, otherwise G=1, -R=1.21 when race is black, otherwise R=1.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Standard Dose EC-MPS | High EC-MPS
Number analyzed (Participants) | 47 | 45
mL/min/1.73m^2
  Baseline (n= 47, 45) | 45.3 (9.5) | 46.4 (11.2)
  Month 3 (n= 44, 43) | 44.6 (10.9) | 48.6 (10.8)
  Change from Baseline to Month 3 (n= 44, 43) | -0.4 (4.6) | 2.1 (4.9)

3. Secondary Outcome: Number of Participants With Treatment Failure Parameters (Biopsy-Proven Acute Rejection (BPAR), Graft Loss, Death, or Loss to Follow-up) at 6 Months
Description: A biopsy-proven acute rejection (BPAR) is defined as a biopsy graded IA, IB, IIA, IIB, or III based on the Banff 1997 classification.The allograft was presumed lost on the day the patient started dialysis and was not able to subsequently be removed from dialysis. If the patient went through a graft nephrectomy, then the day of nephrectomy was the day of graft loss.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Standard Dose EC-MPS | High EC-MPS
Number analyzed (Participants) | 47 | 45
Participants
  Biopsy proven acute rejection | 0 | 0
  Treated acute rejection | 0 | 0
  Graft loss | 0 | 0
  Death | 0 | 0

4. Secondary Outcome: Number of Participants With Graft and Patient Survivals at 6 Months
Description: Graft survival was defined as the number of patients with no graft loss. The allograft was presumed lost on the day the patient started dialysis and was not able to subsequently be removed from dialysis. If the patient went through a graft nephrectomy, then the day of nephrectomy was the day of graft loss. Patient survival was defined as the number of patients alive with or without a functioning graft.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Standard Dose EC-MPS | High EC-MPS
Number analyzed (Participants) | 47 | 45
Participants
  Graft survival | 47 | 45
  Patient survival | 47 | 45

ADVERSE EVENTS:
Time Frame: 6 months
Description: Safety population
Arm/Group | Standard Dose EC-MPS | High EC-MPS
Serious Adverse Events (participants affected / at risk) | 8/47 | 7/45
Other Adverse Events (participants affected / at risk) | 4/47 | 10/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose EC-MPS (N=47) | High EC-MPS (N=45)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Pneumocystis jiroveci infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose EC-MPS (N=47) | High EC-MPS (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.